CLINICAL TRIAL: NCT04413760
Title: Physiological and Psychological Strain in Elementary School Teacher
Acronym: BelaPrim
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Collaborators: Private University of Education Diocese of Linz (Unknown); eduResearch - Upper Austrian Centre for Education Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: A-2018-013
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Work-Related Musculoskeletal Disorders; Work-Related Stress Disorders
Keywords: Musculoskeletal Pain; Psychological Stress; Primary School teachers
MeSH Terms: conditions — Musculoskeletal Pain; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survey will enquire the physical and psychological conditions in primary school teachers in Upper Austria. All primary teachers of the 553 Upper Austrian elementary schools (approximately 5105 persons) will be interviewed between November 2018 and April 2019. The main outcomes will be Musculoskeletal pains in nine body regions, the physical activity and the psychological stress with the "Work-related Behaviour and Experience Patterns" and big five personality traits.

DETAILED DESCRIPTION:
Background: Musculoskeletal disorders (MSD) are the leading cause of pain and loss of function, and are complex complaints of high prevalence, resulting in high costs and the psychosocial disadvantages of these patients. The prevalence of work-related physical stress in primary school teachers worldwide depending on the region ranges from 32% to 67%. Schoolteachers also represent an occupation group among which there appears to be a high prevalence of MSD. Many studies have shown that musculoskeletal pain (MSP) impairs quality of life (QoL) to a varying extent. For working populations, musculoskeletal disorders (MSDs) are considered as being responsible for a substantial impact on QoL and incurring a major economic burden in compensation costs and lost wages. Since being a reason for seeking healthcare, MSDs decrease productivity at work, cause absence due to sickness and even to early retirement.

Musculoskeletal pains top the list of the most common work-related ailments in Austria. In 2018, they were the third-leading cause for taking sick leave. MSD is one of the leading causes of ill-health retirement among schoolteachers. Gender, age, length of employment and awkward posture are found to be associated with higher MSD prevalence rates among teachers. Primary School teachers spend 25% of time in squatting, kneeling, or sitting position on the floor. An additional 26% of their time was spent sitting on small, child-sized furniture. 18% of teachers' activities were involved in flexing at the trunk greater than 20°. Classroom is configured for primary school pupils. The intensity and frequency correlated with ergonomic factors in the work environment.

Beside physical pressures in teachers work, the occupational engagement and individual coping capacity are very important. Schaarschmidt and Kieschke found four types of work-related coping behaviours. These types include psychological aspects of the health. Particular attention is paid to the question of personality factors that facilitate a health-promoting approach to the demands of the profession. The picture for teachers is quite problematic. The teaching profession appears to be associated with higher health risks than other fields of employment. Furthermore, striking gender differences were observed. Female teachers apparently suffer from greater stress than their male colleagues. On the other hand, there are hardly any school-specific or regional differences. Personality traits that prove beneficial for the teaching profession are, in particular, conscientiousness, extraversion and psychological stability. Increased neuroticism is a risk factor for experiencing professional stress and burnout. A low level of neuroticism is a favorable personal disposition in the teaching profession, since everyday teaching is characterized by diverse and permanent social interactions. Therefore, teachers should be expressive, enjoy communicating, be confident, and assertive in socio-communicative situations. In addition, appreciative behavior, friendliness and empathy, team and problem-solving skills are advantageous for teachers.

Schaarschmidt was able to show by coping patterns that in the context of school in Germany and Austria there is a critical distribution of these coping patterns regardless of the type of school. In all school types, at least 50% of the teachers are in the risk patterns (overload, burn-out) and just under 20% are in the healthy pattern, in which there is sufficient positive experience of work, commitment and resilience to the challenges of the profession. This picture becomes even more problematic when one compares the pattern distribution between female and male teachers. A shift to the disadvantage of female teachers is evident in all school types.

Both, musculoskeletal pains and psychological stress, has a great influence on the health and quality of life of primary school teachers.

Aim: The primary aim of this observational study is to enquire the physical and psychological conditions in primary school teachers in Upper Austria. The second goal is to evaluate the influence of physical activity and personal factors on physical and mental health. The personal feedback will evaluate qualitatively in the sense of a holistic view. The authors hope that the results will provide new insights into the factors influencing the works of primary school teachers.

Methods: The survey will conduct by an online questionnaire using the "Questback Enterprise Feedback Suite" tool. The questionnaire included four sections. After the introduction page, followed the physical stress examination with the Nordic Musculoskeletal Questionnaire (NMQ). The second part will survey the psychological stress with the 11 item short test with the "Work-related Behaviour and Experience Patterns" (AVEM) and Big5 personality questionnaire (TIPI G). At third sections, the physical activity level will enquiry with the Short-Version of the International Physical Activity Questionnaire (IPAQ). The demographic characteristics (gender and age) and the risk factors (smoker/non-smoker, teaching profile, Job category and anthropometric parameter) will collect finally.

ELIGIBILITY:
Inclusion Criteria:

All primary schoolteachers in active service at elementary schools in Upper Austria will be included

Exclusion Criteria:

* on maternity leave
* ill-health retirement

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary schoolteachers of all gender, between 21 and 65 year of age, working active at elementary schools in Upper Austria
Sampling Method: Non-Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Level of physical activity | at one point (baseline)
  The physical activity (PA) of the participants was assessed through the German version of the International Physical Activity Questionnaire -Short Form (IPAQ-SF), which includes 6 questions searching the frequency (days per week) and duration (hours) of walking, as well as the intensity of physical activity in the last seven days. The IPAQ calculates the metabolic equivalent (MET) score by asking participants the days and minutes exercised in three categories of intensity (vigorous, moderate, and walking) during the previous one week. The following formula is used to calculate the MET: MET = 8 (vigorous activity)*(minutes) + 4 (moderate activity)*(minutes) +3.3 (walking activity)*(minutes).
Measure stress-related work behaviour | at one point (baseline)
  Work-related Behaviour and Experience Patterns ("Arbeitsbezogenes Verhaltens- und Erlebensmuster" - AVEM) short test using a five-point answer scale to measure the three Dimensions Engagement, Resilience and Emotions. The 5-point Likert scales ranging from 1 (strongly disagree) to 5 (strongly agree). The points if the three Dimensions are assigned to the 2 patterns G ("Health") and S ("Unambitious") or the risk pattern A ("Overexertion") and B ("Burnout"). The higher percentage distribution on the patterns G and S is better, more points for the risk patterns A and B shows a poorer mental health.
Prevalence of pain in nine region of the body with the Nordic Musculoskeletal Questionnaire (NMQ) | at one point (baseline)
  The Questionnaire evaluating the prevalence of pain (dichotomous scale, "yes" or "no") in the neck, shoulders, upper back, elbows, lower back, wrists/hands, hips/thighs, knees and ankles/feet at the last week and at the last 12 months. The prevalence can reach from 0% (no participant answered "yes") to 100% (all participants answered "yes").
Intensity of pain in nine region of the body with the Visual Analogue Scale (VAS) | at one point (baseline)
  Subjects will report their pain intensity in the neck, shoulders, upper back, elbows, lower back, wrists/hands, hips/thighs, knees and ankles/feet at the last week and at the last 12 months by means of VAS. The VAS used for this study ranges from 0 (no pain) to 10 (heavy pain) points.

SECONDARY OUTCOMES:
Big Five personality traits | at one point (baseline)
  The openness, conscientiousness, extraversion, agreeableness and neuroticism will survey at the Trier Integrated Personality Inventory (TIPI). A ten-item measure of the Big Five personality dimensions - 2 items for each of the 5 dimensions. Each item is rated on a 7-point scale that ranges from 1 (disagree strongly) to 7 (agree strongly). The result shows the personal distribution of the personal Big 5 personality traits.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hoppe, MHPE, Principal Investigator — University of Applied Sciences for Health Professions Upper Austria
Locations (1):
- University of Applied Sciences for Health Professions Upper Austria, Linz, Upper Austria, Austria

REFERENCES:
- [Background] Olaya-Contreras P, Styf J. Biopsychosocial function analyses changes the assessment of the ability to work in patients on long-term sick-leave due to chronic musculoskeletal pain: the role of undiagnosed mental health comorbidity. Scand J Public Health. 2013 May;41(3):247-55. doi: 10.1177/1403494812473380. Epub 2013 Jan 29. PMID 23361388
- [Background] Tuzun EH. Quality of life in chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):567-79. doi: 10.1016/j.berh.2007.03.001. PMID 17603000
- [Background] Brown J, Gilmour WH, Macdonald EB. Ill health retirement in Scottish teachers: process, outcomes and re-employment. Int Arch Occup Environ Health. 2006 May;79(5):433-40. doi: 10.1007/s00420-005-0060-9. Epub 2005 Nov 25. PMID 16308706
- [Background] Erick PN, Smith DR. A systematic review of musculoskeletal disorders among school teachers. BMC Musculoskelet Disord. 2011 Nov 17;12:260. doi: 10.1186/1471-2474-12-260. PMID 22087739
- [Background] Maguire M, O'Connell T. Ill-health retirement of schoolteachers in the Republic of Ireland. Occup Med (Lond). 2007 May;57(3):191-3. doi: 10.1093/occmed/kqm001. Epub 2007 Feb 22. PMID 17317705
- [Background] Yue P, Liu F, Li L. Neck/shoulder pain and low back pain among school teachers in China, prevalence and risk factors. BMC Public Health. 2012 Sep 14;12:789. doi: 10.1186/1471-2458-12-789. PMID 22978655
- [Background] Grant KA, Habes DJ, Tepper AL. Work activities and musculoskeletal complaints among preschool workers. Appl Ergon. 1995 Dec;26(6):405-10. doi: 10.1016/0003-6870(95)00057-7. PMID 15677041
- [Background] Slack-Smith LM, Read AW, Darby J, Stanley FJ. Health of caregivers in child care. Child Care Health Dev. 2006 Jan;32(1):111-9. doi: 10.1111/j.1365-2214.2006.00577.x. PMID 16398797
- [Background] Arvidsson I, Gremark Simonsen J, Dahlqvist C, Axmon A, Karlson B, Bjork J, Nordander C. Cross-sectional associations between occupational factors and musculoskeletal pain in women teachers, nurses and sonographers. BMC Musculoskelet Disord. 2016 Jan 18;17:35. doi: 10.1186/s12891-016-0883-4. PMID 26781760
- [Background] Kieschke U, Schaarschmidt U. Professional commitment and health among teachers in Germany: A typological approach. In: Learning and Instruction. 2008; 18 (5): 429-437. DOI: 10.1016/j.learninstruc.2008.06.005.
- [Background] Samad NIA, Abdullah HSM, Tamrin SBM, Hashim Z. Prevalence of Low Back Pain and its Risk Factors among School Teachers. In: American Journal of Applied Sciences. 2010; 7 (5): 634-639. DOI: 10.3844/ajassp.2010.634.639.
- [Background] Horng YS, Hsieh SF, Wu HC, Feng CT, Lin MC. Work-related Musculoskeletal Disorders of the Workers in a Child Care Institution. In: Tw J Phys Med Rehabil. 2008; 36 (1): 15-21.
- [Background] Mayr J. Ein Lehramtsstudium beginnen? Ein Lehramtsstudium beginnen lassen? Laufbahnberatung und Bewerberauswahl konstruktiv gestalten. In: B. Weyand, M. Justus, & M. Schratz (Hg.): Auf unsere Lehrerinnen und Lehrer kommt es an. Geeignete Lehrer/-innen gewinnen, (aus)bilden und fördern. Essen. Stifterverband. 2012; 38-57.
- [Background] Maslach C, Schaufeli WB, Leiter MP. Job burnout. Annu Rev Psychol. 2001;52:397-422. doi: 10.1146/annurev.psych.52.1.397. PMID 11148311
- [Background] Schaarschmidt U. Eignung für den Lehrerberuf frühzeitig erkennen und kontinuierlich fördern. Implikationen aus den Potsdamer Lehrerstudien. In: B. Weyand, M. Justus, & M. Schratz (Hg.): Auf unsere Lehrerinnen und Lehrer kommt es an. Geeignete Lehrer/-innen gewinnen, (aus)bilden und fördern. Essen: Stifterverband. 2012; 58-77.
- [Background] Sliwka A, Klopsch B. Auf den Lehrer/ die Lehrerin kommt es an. Lehrerbildung und Lehrerprofessionalität in internationaler Perspektive. In: B. Weyand, M. Justus, & M. Schratz (Hg.): Auf unsere Lehrerinnen und Lehrer kommt es an. Geeignete Lehrer/-innen gewinnen, (aus)bilden und fördern. Essen: Stifterverband. 2012; 14-35.
- [Background] Schaarschmidt U. Halbtagsjobber? Psychische Gesundheit im Lehrerberuf - Analyse eines veränderungsbedürftigen Zustandes. Weinheim: Beltz. 2004
- [Background] Kieschke U. Arbeit, Persönlichkeit und Gesundheit. Beiträge zu einer differentiellen Psychologie beruflichen Belastungsgeschehens. Berlin: Logos Verlag Berlin. 2003
- [Background] Mayr J. Persönlichkeitsmerkmale und Interessen als Korrelate der Entwicklung, der Kompetenz und des Befindens im Lehrberuf. Habilitation. Universität Lüneburg, Lüneburg. Fachbereich Erziehungswissenschaften. 2001
- [Background] Müller FH, Andreitz I, Hanfstingl B. Die Bedeutung der Selbstbestimmung von Lehrpersonen für Unterricht und Lernen. Empirische Befunde aus dem Interventionsprojekt IMST. Klagenfurt: Eigenverlag IUS 2008
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Gosling, Samuel D.; Rentfrow, Peter J.; Swann, William B. (2003): A very brief measure of the Big-Five personality domains. In: Journal of Research in Personality 37 (6), S. 504-528. DOI: 10.1016/S0092-6566(03)00046-1.
- [Background] Schaarschmidt U. AVEM. - ein persönlichkeitsdiagnostisches Instrument für die berufsbezogene Rehabilitation. In: Psychologische Diagnostik. Vom 18. bis 20. November 2005 im Bildungszentrum Erkner. Unter Mitarbeit von Christine Gerhard. Bonn: Dt. Psychologen-Verl. (Reha-Psychologie, 24.2005). 2006; 59-82.